CLINICAL TRIAL: NCT05712421
Title: A Randomized, Double-blind, Dose-Conversion Study to Evaluate the Safety and Efficacy of Hormone Replacement Therapy With North Star Compared to Levothyroxine in Subjects With Primary Hypothyroidism Who Are Euthyroid on Levothyroxine Replacement Therapy
Brief Title: A Study Evaluation the Safety and Efficacy of Hormone Replacement Therapy With North Star Compared to Levothyroxine in Patients With Primary Hypothyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuvosyn Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NorthStar-02-001
Record Dates: First submitted 2023-01-18; First posted 2023-02-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- North Star (Experimental)
  Interventions: Drug: North Star
- Levothyroxine (Active Comparator)
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: North Star — North Star
  Arms: North Star
Drug: Levothyroxine — Levothyroxine
  Arms: Levothyroxine

SUMMARY:
The North Star study is a multi-center, Phase 2, double-blind, randomized, parallel group clinical study to evaluate the safe and effective dose conversion from Levothyroxine to North Star therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary hypothyroidism
* On continuous thyroid replacement therapy for at least 6 months before Study Entry
* On a stable daily dose of LT4 for a minimum of 12 weeks prior to Screening
* Agree to practice a method of contraception
* Female patients not pregnant or lactating at Screening
* Agree to practice a method of contraception of greater than 90% reliability
* Willing to give written informed consent for the Study
* Provide written authorization for use and disclosure of protected health information

Exclusion Criteria:

* Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation or excretion of North Star or levothyroxine
* Hospitalization for a major illness within 4 weeks prior to Screening
* Anticipated initiation or change in concomitant medications
* Concomitant use of prohibited medications or supplements
* Participated in another investigational new drug study within 30 days or 5 half-lives of the IMP, whichever is longer, prior to the first study drug administration.
* For female subjects, be pregnant, nursing or planning to become pregnant during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
The ratio of the LT4 dose (mcg/day) at screening to North Star (mg/day) at the end of the treatment period required to achieve and maintain serum thyroid-stimulating hormone (TSH) levels within the normal reference range. | Week 30

SECONDARY OUTCOMES:
Proportion of subjects who are euthyroid as determined by serum TSH level within the normal reference range at the end of the treatment period. | Week 30

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Neuvosyn Investigational Site, Birmingham, Alabama
  - Neuvosyn Investigational Site, Canoga Park, California
  - Neuvosyn Investigational Site, Greenbrae, California
  - Neuvosyn Investigational Site, Toluca Lake, California
  - Neuvosyn Investigational Site, Farmington, Connecticut
  - Neuvosyn Investigational Site, Boca Raton, Florida
  - Neuvosyn Investigational Site, Miami, Florida
  - Neuvosyn Investigational Site, Sunrise, Florida
  - Neuvosyn Investigational Site, Acworth, Georgia
  - Neuvosyn Investigational Site, Atlanta, Georgia
  - Neuvosyn Investigational Site, Columbus, Georgia
  - Neuvosyn Investigational Site, Sugar Hill, Georgia
  - Neuvosyn Investigational Site, Saginaw, Michigan
  - Neuvosyn Investigational Site, Gladstone, Missouri
  - Neuvosyn Investigational Site, Williamsville, New York
  - Neuvosyn Investigational Site, Denver, North Carolina
  - Neuvosyn Investigational Site, Winston-Salem, North Carolina
  - Neuvosyn Investigational Site, Beavercreek, Ohio
  - Neuvosyn Investigational Site, Columbus, Ohio
  - Neuvosyn Investigational Site, Georgetown, Texas
  - Neuvosyn Investigational Site, Houston, Texas
  - Neuvosyn Investigational Site, Katy, Texas
  - Neuvosyn Investigational Site, Lewisville, Texas
  - Neuvosyn Investigational Site, Paris, Texas
  - Neuvosyn Investigational Site, Pearland, Texas
  - Neuvosyn Investigational Site, Stafford, Texas

IPD SHARING:
Plan to Share IPD: No